CLINICAL TRIAL: NCT02622282
Title: Text Messaging to Promote Walking Among Latino Adults at Risk for PAD
Brief Title: Text Messaging to Promote Walking Among Latino Adults at Risk for Peripheral Arterial Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00003190; R56AG047590 (NIH)
Record Dates: First submitted 2015-12-02; First posted 2015-12-04 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Peripheral Arterial Disease
Keywords: physical activity; physical inactivity; PAD; Diabetes; High blood pressure; High cholesterol; Smoking
MeSH Terms: conditions — Peripheral Arterial Disease; Motor Activity; Sedentary Behavior; Diabetes Mellitus; Hypertension; Hypercholesterolemia; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (Experimental): Participants will receive text messages and telephone calls during the length of their participation. Participants will receive a handout with information on PAD and physical activity.
  Interventions: Other: Text Messages; Other: Phone Calls; Other: Handout
- Control Group (Active Comparator): Participants will receive a handout with information on PAD and physical activity.
  Interventions: Other: Handout

INTERVENTIONS:
Other: Text Messages — Text messages will be sent one time per day. Text messages will include messages to motivate and inform participants on the importance of walking.
  Arms: Experimental Group
Other: Phone Calls — Participants may receive a telephone call every two weeks for one month followed by once per month for two months.
  Arms: Experimental Group
Other: Handout — Handout includes information specific to participant's condition and ways to promote an active lifestyle.

SUMMARY:
The purpose of this study is to learn about the impact of text messaging on physical activity in persons with risk factors for peripheral arterial disease (PAD).

DETAILED DESCRIPTION:
Thirty-five million Latinos live in the U.S. and nearly 14% have peripheral arterial disease (PAD) defined as a build-up of plaque in the arteries that supply blood to the legs. Approximately 40% have at least one risk for PAD (i.e., aged 70 years and older, diabetes, high blood pressure, high blood cholesterol, or smoking). Persons with at least one risk factor and who are physically inactive are more likely to suffer from severe PAD. Physical inactivity is highly prevalent in Latinos and a major risk factor for PAD. Physical inactivity affects 50% of Latinos aged 60 years and older.

Participation in this study will last for about 3 months. Participants will be randomized to one of two groups. One group will receive text messages, brief telephone calls, and a handout. The other group will only receive the handout. The study will be looking at how the different groups respond to the different interventions used in the study.

ELIGIBILITY:
Inclusion Criteria:

* Latino adults
* English or Spanish speaking
* Have one or more of the following: diabetes mellitus, smoking, hypertension, or hyperlipidemia.
* Adults age 70 years or older, regardless of having one or more the above noted risk factors for PAD, will also be eligible for enrollment.

Exclusion Criteria:

* Pregnancy
* Prior major amputation (foot or lower leg) or critical leg ischemia (tissue loss, gangrene, or ulcers)
* Use of supplemental oxygen
* Myocardial infarction within preceding 3 months

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2016-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in Physical Activity | Change from Baseline to 3 Months
  All participants will use a pedometer. Mean change will be measured based on steps per day.

SECONDARY OUTCOMES:
Change in Exercise Behavior | Change from Baseline to 3 Months
  Change will be measured using the Exercise Behaviors Survey.
Change in Quality of Life | Change from Baseline to 3 Months
  Change will be measured using the Medical Outcomes Study (MOS) Short Form 36. The survey has 36 questions. Scores are coded based on response by participant. A score of 100 indicates the most favorable situation while a score of 0 would indicate the least favorable.

CONTACTS AND LOCATIONS:
Overall Officials: Tracie C. Collins, MD, MPH, Principal Investigator — University of Kansas Medical Center
Locations (1):
- KU School of Medicine - Wichita, Wichita, Kansas, United States

REFERENCES:
- [Derived] Collins TC, Lu L, Valverde MG, Silva MX, Parra-Medina D. Efficacy of a multi-component intervention to promote physical activity among Latino adults: A randomized controlled trial. Prev Med Rep. 2019 Aug 7;16:100965. doi: 10.1016/j.pmedr.2019.100965. eCollection 2019 Dec. PMID 31453076